CLINICAL TRIAL: NCT04141176
Title: Evaluation of the Efficacy of Sleepinnov© (Spiri+) Continuous Positive Airway Pressure Device
Brief Title: Obstructive Sleep Apnea Syndrome: Evaluation of the Efficacy of Sleepinnov© (Spiri+) Continuous Positive Airway Pressure Device
Acronym: Spiri+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sleepinnov Technology (Industry)
Collaborators: University Hospital, Grenoble (Other); ICUREsearch (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-A03014-51
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2019-11

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Continuous positive airway pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: It's a prospective, open, monocentric study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spiri+ (Experimental): new CPAP device
  Interventions: Device: Spiri+

INTERVENTIONS:
Device: Spiri+ — CPAP Spiri+ will be weared during one night for each included patient.The validation of the CPAP Spiri+ algorithm will be in the first 10 patients and appreciation of overall clinical efficacy on the 10 last OSAS.

SUMMARY:
Continuous Positive Airway Pressure (CPAP) is the reference treatment of patients suffering from Obstructive Sleep Apnea Syndrome (OSAS).This device functions as a pneumatic stent that stabilizes the upper airway, prevents periodic collapses during sleep.The correction of abnormal respiratory events during sleep allows improvement of symptoms related to OSAS and restores quality of life.The purpose of this study is to validate the efficacy of a new CPAP brand developed by Sleepinnov©.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) is characterized by the repetitive occurrence of partial or complete pharyngeal obstructions during sleep.Continuous Positive Airway Pressure (CPAP) is the first line treatment of OSAS.

The aim of the prospective monocentric two steps pilot study SPIRI+ is to validate the efficacy of a new CPAP brand developed by Sleepinnov©.

* the first step will validate the capability of the algorithm to appropriately detect of abnormal repiratory events during sleep.the metrics will be a comparison of the total number of events detected by the CPAP Sleepinnov© with data arising from a concurrent polysomnography.
* the second step will check overall clinical efficacy of the new CPAP device by assessing the percentage of OSAS with an index of residual events below 10 and 5 per hour.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed and untreated Obstructive sleep apnea syndrome (IAH >15/hour) with an indication of treatment with CPAP
* Patients who have given their informed written consent

Exclusion Criteria:

* Pregnant or lactating women
* Patients not affiliated to the French social security system or equivalent
* Patient deprived of liberty by judicial or administrative decision
* Patients under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-11-16 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
Part 1: Validation of algorithm detection of respiratory events | baseline
  Comparison of the total number of events detected by the CPAP Sleepinnov© with data arising from a concurrent polysomnography.
Part 2: Validation of overall clinical efficacy | baseline
  Percentage of OSAS with an index of residual events below 10 and 5 per hour

SECONDARY OUTCOMES:
Part 1: | baseline
  Compare the different types of events detected by the Spiri + CPAP algorithm to the concomitant respective indices scored during concurrent

CONTACTS AND LOCATIONS:
Overall Officials: Renaud Tamisier, PhD, Principal Investigator — University Hospital, Grenoble; Jean-Louis Pépin, PhD, Principal Investigator — University Hospital, Grenoble; Marie Destors, MD, Principal Investigator — University Hospital, Grenoble; Sébastien Baillieul, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, La Tronche, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Senaratna CV, Perret JL, Lodge CJ, Lowe AJ, Campbell BE, Matheson MC, Hamilton GS, Dharmage SC. Prevalence of obstructive sleep apnea in the general population: A systematic review. Sleep Med Rev. 2017 Aug;34:70-81. doi: 10.1016/j.smrv.2016.07.002. Epub 2016 Jul 18. PMID 27568340
- [Background] Levy P, Kohler M, McNicholas WT, Barbe F, McEvoy RD, Somers VK, Lavie L, Pepin JL. Obstructive sleep apnoea syndrome. Nat Rev Dis Primers. 2015 Jun 25;1:15015. doi: 10.1038/nrdp.2015.15. PMID 27188535